CLINICAL TRIAL: NCT01435499
Title: A Feasibility and Toxicity Study of a Granulocyte-Macrophage Colony-Stimulating Factor (GM-CSF) Secreting Allogeneic Melanoma Vaccine Administered Alone or in Combination With Cyclophosphamide in Subjects With Surgically Resected At-Risk Melanoma
Brief Title: Safety Study of a Melanoma Vaccine (GVAX) With or Without Cyclophosphamide in Patients With Surgically Resected Melanoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: The John P. Hussman Foundation (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: J1112
Record Dates: First submitted 2011-09-08; First posted 2011-09-16 (Estimated); Last update posted 2016-05-24 (Estimated); Status verified 2016-05

CONDITIONS: Melanoma
Keywords: immunotherapy; vaccine; GVAX; GM-CSF
MeSH Terms: conditions — Melanoma | interventions — Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Cohort A (Experimental): Cohort A will receive four doses of vaccine, each containing 5E7 melanoma GVAX cells.
  Interventions: Biological: melanoma GVAX
- Cohort B (Experimental): Cohort B will receive four doses of vaccine, each containing 2E8 melanoma GVAX cells.
  Interventions: Biological: melanoma GVAX
- Cohort C (Experimental): Cohort C will receive four doses of vaccine, each containing 2E8 melanoma GVAX cells. One day prior to each vaccination, patients in cohort C will receive a single, low dose of intravenous cyclophosphamide.
  Interventions: Biological: melanoma GVAX; Drug: Cyclophosphamide

INTERVENTIONS:
Biological: melanoma GVAX — Melanoma GVAX is given as intradermal injections every 28 days x 4 doses. Cohort A will receive 5E7 cells/dose; cohorts B and C will receive 2E8 cells/dose.
Drug: Cyclophosphamide — 200mg/m2 given as a single dose, intravenously, one day prior to each of the 4 vaccinations to patients in cohort C only
  Arms: Cohort C

SUMMARY:
The primary objective of this study is to evaluate the safety and feasibility of administering an allogeneic GM-CSF-secreting lethally irradiated whole melanoma cell vaccine ("melanoma GVAX"), alone or in combination with low dose cyclophosphamide (CPM), for the adjuvant treatment of patients with surgically resected stage IIB-IV melanoma. Secondarily, the investigators will assess in vitro correlates of anti-melanoma immunization by melanoma GVAX, including serological and cellular immune responses in patients treated with either the vaccine alone or the vaccine given with low dose CPM.

ELIGIBILITY:
Inclusion Criteria:

* Any patient age ≥18 years with melanoma of cutaneous or mucosal origin, and with clinicopathologic stage IIB, IIC, III or IV that has been completely resected
* Patients must be able to provide informed consent.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
* Life expectancy of at least 6 months.
* Adequate hematologic function.
* Adequate renal function
* Adequate hepatic function
* Patients of both genders must agree to practice effective birth control during the study period and for at least 4 weeks after the last treatment.

Exclusion Criteria:

* Patients whose primary site of melanoma is ocular.
* Are undergoing or have undergone in the past 4 weeks any systemic treatment for melanoma.
* Are undergoing or have undergone in the past 2 weeks any surgery or focal radiation therapy.
* Have active systemic infections, coagulation disorders (including therapeutic anticoagulation), or other major medical or psychiatric illnesses.
* Are known to be positive for hepatitis B surface antigen, anti-Hepatitis C Virus or anti-Human Immunodeficiency Virus (HIV) antibody (because of possible immune effects of these conditions).
* Documented history of autoimmune disease, for example, systemic lupus erythematosus, sarcoidosis, rheumatoid arthritis, glomerulonephritis, or vasculitis.
* Any form of primary or secondary immunodeficiency. This would include hereditary disorders such as ataxia-telangiectasia or Wiskott-Aldrich syndrome, or acquired immune deficiencies such as following bone marrow transplantation.
* Requirement for systemic steroid therapy or immunosuppressive therapy.
* Have received any type of cancer immunotherapy, including but not limited to interleukin-2, interferon alfa or melanoma vaccines.
* Have been diagnosed with another invasive cancer within the past 3 years.
* Radiographic evidence of melanoma recurrence.
* Pregnant or lactating women.
* Known or suspected hypersensitivity to GM-CSF, pentastarch, hetastarch, corn, Dimethyl sulfoxide, fetal bovine serum or trypsin (porcine origin).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2011-09; Primary Completion 2013-01 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events as a Measure of Safety and Tolerability of Administering Melanoma GVAX With and Without Cyclophosphamide | 2.5 years
  To determine the side effects and tolerability of administering an allogeneic GM-CSF-secreting lethally irradiated whole melanoma cell vaccine ("melanoma GVAX"), alone or in combination with low dose cyclophosphamide, for the adjuvant treatment of patients with surgically resected stage IIB-IV melanoma.

SECONDARY OUTCOMES:
In vitro correlates of anti-melanoma immunization | 2.5 Years
  We will assess in vitro correlates of anti-melanoma immunization by melanoma GVAX, including serological and cellular immune responses in patients treated with either the vaccine alone or the vaccine given with low dose cyclophosphamide. These investigations are exploratory in nature and will not affect clinical care.

CONTACTS AND LOCATIONS:
Overall Officials: Evan J Lipson, M.D., Principal Investigator — The Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins
Locations (1):
- The Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland, United States

REFERENCES:
- [Derived] Lipson EJ, Sharfman WH, Chen S, McMiller TL, Pritchard TS, Salas JT, Sartorius-Mergenthaler S, Freed I, Ravi S, Wang H, Luber B, Sproul JD, Taube JM, Pardoll DM, Topalian SL. Safety and immunologic correlates of Melanoma GVAX, a GM-CSF secreting allogeneic melanoma cell vaccine administered in the adjuvant setting. J Transl Med. 2015 Jul 5;13:214. doi: 10.1186/s12967-015-0572-3. PMID 26143264